CLINICAL TRIAL: NCT07166081
Title: A Phase 1, Double-Blind, Randomized, Ascending-Dose, Placebo-Controlled, Multiple-dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of BGM0504 Tablets Orally Administered in Non-diabetic Overweight or Obese Adult Subjects
Brief Title: Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of BGM0504 Tablets in Non-diabetic Overweight or Obese Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM0504 Oral-P1-CPK01-US
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Non-diabetic Overweight or Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 20 mg BGM0504 administered orally
  Interventions: Drug: BGM0504
- Cohort 2 (Experimental): 40 mg BGM0504 administered orally
  Interventions: Drug: BGM0504
- Cohort 3 (Experimental): 60 mg BGM0504 administered orally
  Interventions: Drug: BGM0504
- Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo
- Cohort 4 (Experimental): 80mg BGM0504 administered orally
  Interventions: Drug: BGM0504

INTERVENTIONS:
Drug: BGM0504 — Administered orally
  Arms: Cohort 1
Drug: BGM0504 — Administered orally
  Arms: Cohort 2
Drug: BGM0504 — Administered orally
  Arms: Cohort 3
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: BGM0504 — Administered orally
  Arms: Cohort 4

SUMMARY:
This is a Phase 1, single-center, randomized, placebo-controlled, ascending dose study. The study will evaluate the pharmacokinetics (PK), pharmacodynamic (PD), preliminary efficacy, safety and tolerability of BGM0504 following daily oral administrations in non-diabetic overweight or obese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) meeting one of the following requirements:

  1. Between ≥ 30.0 kg/m2 and ≤ 40.0 kg/m2 (obese); OR
  2. Between ≥ 27.0 kg/m2 and < 30.0 kg/m2 (overweight) with at least 1 of the following: One or more symptoms of prediabetes (impaired fasting plasma glucose and/or abnormal glucose tolerance), grade 1 hypertension, simple fatty liver or dyslipidemia
* Have a stable body weight (<5% self-reported change during the previous 12 weeks) before screening
* Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the schedule, requirements and restrictions of the study.

Exclusion Criteria:

* Have allergic predisposition (allergic to 3 or more foods or drugs), or are allergic to glucagon-like peptide-1 (GLP-1) receptor agonists or suffer from severe allergic diseases (asthma, urticaria, eczematous dermatitis).
* Have received GLP-1 receptor agonists or similar drugs containing the same target within 12 weeks before screening.
* Have received drugs that have an impact on body weight within 12 weeks before screening.
* Known type I/II diabetes.
* History of acute or chronic pancreatitis or pancreatic injury.
* History of drug abuse or alcoholism at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Number of treatment adverse events | 11 weeks
  The relationship of each adverse event tothe investigational product was assessed by the investigator

SECONDARY OUTCOMES:
Pharmacokinetic endpoint: Concentration of BGM0504 in plasma | 11 weeks
Change in fasting weight at week 11 | 11 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Inc, Baltimore, Maryland, United States